CLINICAL TRIAL: NCT04375657
Title: Thymus Regeneration, Immunorestoration, and Insulin Mitigation Extension Trial
Acronym: TRIIM-X
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intervene Immune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRIIM-X
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Epigenetic Aging; Immunosenescence

STUDY DESIGN:
Intervention Model Description: TRIIM-X is an expanded pilot clinical study that will evaluate a personalized combination treatment regimen for thymus regeneration.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRIIM Treatment (Experimental)
  Interventions: Combination Product: TRIIM Treatment
- Active Control (Active Comparator)
  Interventions: Combination Product: Active Control

INTERVENTIONS:
Combination Product: TRIIM Treatment — Personalized combination of somatropin, metformin, and DHEA
  Arms: TRIIM Treatment
Combination Product: Active Control — Metformin and DHEA
  Arms: Active Control

SUMMARY:
The TRIIM-X trial is an expanded pilot clinical study that will evaluate a personalized combination treatment regimen for thymus regeneration. The thymus is a part of the immune system that declines markedly with age, and regenerating it may prevent or reverse key aspects of immunosenescence (immune system aging) and potentially prevent or reverse key parts of the aging process more generally. The study will evaluate biomarkers for epigenetic aging and immunosenescence, as well as evaluate established clinical measures and risk factors for prevention of physical frailty, cancer, cardiovascular disease, diabetes, dementia, and also infectious diseases, including flu and COVID-19.

The study uses multiple agents in combination with personalized doses of recombinant human growth hormone (somatropin), metformin, and DHEA, in a similar manner to how the combination treatment was applied in the earlier TRIIM trial at Stanford, which demonstrated strong statistical significance for the primary efficacy endpoints that will be evaluated in TRIIM-X. Somatropin is approved by the FDA for adult growth hormone deficiency and its use in the study is guided by prior safety data established for that use and also based on safety data available on its prior use in the TRIIM trial and in clinical practice in healthy elderly individuals. There will also be control groups that enable testing of biomarker variability and the contribution of individual medications within the combination treatment.

The objective of the study is to obtain information needed for designing an effective personalized and adaptive treatment regimen for a larger and more diverse study population, and to obtain additional proof of principle for the new use of the medications and biomarkers for preventive medicine. The duration of treatment in the TRIIM-X trial will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers
* Aged 40 to 80 years, inclusive
* All ethnicities
* Able to participate in 12-month study
* Able to provide informed consent

Exclusion Criteria:

* Malignancies or high risk of malignancy, as suggested by familial risk or personal medical history
* Premenopausal women
* Postmenopausal women on HRT
* IGF-1 levels < 90 ng/ml or >300 ng/ml
* Diagnosed or suspected growth hormone resistance
* Known growth hormone deficiency based on stimulation testing
* Pre-existing carpal tunnel syndrome
* Significant arthritis/arthralgia/joint swelling
* Bradycardia (<55 bpm), significant hypertension (systolic >160 mmHg, or diastolic >90 mmHg) despite treatment, serious angina, or other serious cardiovascular disease or cardiovascular disease risk factors
* Excessive skin growths (e.g., flat warts) without cryosurgical options
* BMI of 35 or greater
* PSA level above the age-adjusted normal range for reasons other than confirmed prostatitis
* Testosterone levels above the upper limit of normal
* Levels of C-reactive protein (CRP) above the upper limit of normal
* Type 1 or pre-existing Type 2 diabetes
* Uncorrected hypothyroidism
* HIV infection
* Allergy or other sensitivity to study medications
* Other unstable medical conditions
* Use of GH within the last 5 years
* Participation in a clinical research trial within 30 days prior to enrollment
* Use of chronic glucocorticoid therapy
* Unwilling to discontinue androgen supplementation if testosterone levels are above the upper limit of normal
* Ongoing treatment with carbonic anhydrase inhibitors
* Ketogenic diet, calorie-restricted diet, or prolonged fasting, without willingness to discontinue these diets or adhere to an alternative diet during the study
* Alcoholism or drug addiction
* Smoking or unwillingness to quit smoking
* Cognitive impairment, illiteracy, inability or unwillingness to give voluntary informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age | 12 months
  DNA methylation based epigenetic age (GrimAge)
Thymus Regeneration | 12 months
  Thymic density based on MRI or CT
Safety and Tolerability | 12 months
  Incidence of treatment-related adverse effects

SECONDARY OUTCOMES:
Immunosenescence | 12 months
  Assessment of naive T cells and immune cell function

CONTACTS AND LOCATIONS:
Locations (1):
- Intervene Immune, Torrance, California, United States

REFERENCES:
- [Background] Fahy GM, Brooke RT, Watson JP, Good Z, Vasanawala SS, Maecker H, Leipold MD, Lin DTS, Kobor MS, Horvath S. Reversal of epigenetic aging and immunosenescent trends in humans. Aging Cell. 2019 Dec;18(6):e13028. doi: 10.1111/acel.13028. Epub 2019 Sep 8. PMID 31496122